CLINICAL TRIAL: NCT03685851
Title: Post Operative Visual Acuity for Descemet Stripping Automated Endothelial Keratoplasty (DSAEK) and UT-DSAEK
Brief Title: Post Operative Visual Acuity for DSAEK and UT-DSAEK
Acronym: POVIAD
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-04Obs-CHRMT
Record Dates: First submitted 2018-09-25; First posted 2018-09-26 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-09

CONDITIONS: Corneal Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- UT-DSAEK: With graft 6 months thick less than 100 µm
  Interventions: Procedure: DSAEK type corneal transplant
- DSAEK: With graft thicker than 100 µm
  Interventions: Procedure: DSAEK type corneal transplant

INTERVENTIONS:
Procedure: DSAEK type corneal transplant — All surgeries were performed by the same surgeon and according to the same protocol

SUMMARY:
To study the correlation between graft size in DSAEK (Descemet Stripping Automated Endothelial Keratoplasty) and UT (ultra thin)-DSAEK type corneal transplants to the visual acuity 6 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent DSAEK surgery
* Patients in department of ophthalmology between february 2012 and june 2017

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent DSAEK surgery between february 2012 and june 2017
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2015-04-01 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Postoperative visual acuity | Month 6
  postoperative visual acuity in logmar

SECONDARY OUTCOMES:
Pachymetry | Month 6
  Measurement of the thickness of the cornea